CLINICAL TRIAL: NCT01149070
Title: An Observational Program to Evaluate Efficacy, Safety and Clinical Outcomes of Currently Used Pharmaceutical Therapies for Controlled Ovarian Stimulation (COS) in Assisted Reproductive Techniques (ART)
Brief Title: An Observational Study to Evaluate Efficacy, Safety and Clinical Outcomes of Currently Used Pharmaceutical Therapies for Controlled Ovarian Stimulation in Assisted Reproductive Techniques
Acronym: ESCORT
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Kft., Hungary (Industry)
Responsible Party: Sponsor
Other Study IDs: 700623-506
Record Dates: First submitted 2010-05-28; First posted 2010-06-23 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Infertility
Keywords: Infertility; Controlled ovarian stimulation; Reproductive techniques, assisted; Sperm injections, intracytoplasmic; Gonal-f; Ovitrelle
MeSH Terms: conditions — Infertility; Helping Behavior

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
Human gonadotrophins have been successfully used for the treatment of infertility for more than 30 years. This observational study is being conducted to evaluate the efficacy and safety of the gonadotropins used for controlled ovarian stimulation (COS) in assisted reproductive technologies (ART).

DETAILED DESCRIPTION:
The objective of this observational program is to evaluate the efficacy and safety of the gonadotropins used for COS in ART. The clinical use of the various progesterone preparations will also be monitored and registered. All medications will be used according to normal clinical practice, as described in the Summary of Product Characteristics (SmPC). From the start of the program cycles data will be collected prospectively for 12 months and also a substantial amount of cycles will be analyzed retrospectively for the previous 6 months. Data will be collected from all subjects stimulated by follicle stimulating hormone (FSH), with or without down regulation and exogenous lutenizing hormone (LH) supplementation, and final follicular maturation triggered by human chorionic gonadotropin (hCG) and luteal phase support by any means for COS in ART and intracytosolic sperm injection (ICSI). All the medications should be used according to usual clinical practice. Data related to pretreatment (basal examination, history of infertility, LH suppression), stimulation (gonadotropin use, concomitant medications, luteal phase supplementation, ovulation triggering, cycle cancellation, fertilization methods), safety aspects and clinical outcome will be captured.

ELIGIBILITY:
Inclusion Criteria:

* This is a registry wherein data will be collected from all subjects stimulated by FSH, with- or without down regulation and exogenous luteinising hormone (LH) supplementation, and final follicular maturation triggered by hCG and luteal phase support by any means for controlled ovarian stimulation (COS) in assisted reproductive technique (ART) and intracytoplasmic sperm injection (ICSI).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects undergoing ART
Sampling Method: Non-Probability Sample
Enrollment: 10103 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of gonadotropins will be assessed by pregnancy outcome | From the start of the program cycles up to 12 months (data will be collected prospectively for 12 months and also a substantial amount of cycles will be analyzed retrospectively for the previous 6 months)
  Duration and dose of gonadotropin; ovulation triggering; cycle cancellation reasons; clinical pregnancy at week 8; gestational sac size; foetal heart beat; ectopic pregnancy; early pregnancy loss; ongoing pregnancy with fresh and frozen embryos; pregnancy outcome (number, weight, length and percentile of born children); endometrial thickness; number of oocytes per retrieval; size of leading follicle; number of oocytes fertilized; total number of embryos; number of fresh embryos transferred; fertilization rate; number of cryopreserved embryos per FET; mean quality score of transferred embryos.
Safety assessments include recording of adverse events (AEs), serious adverse events (SAEs), AE resulting in cancellation, drug related AEs, ovarian hyperstimulation syndrome [OHSS (mild, moderate, severe, none)]. | From the start of the program cycles up to 12 months (data will be collected prospectively for 12 months and also a substantial amount of cycles will be analyzed retrospectively for the previous 6 months)

SECONDARY OUTCOMES:
Clinical outcomes of the various progesterone preparations will be monitored and registered by assessing clinical pregnancy | From the start of the program cycles up to 12 months (data will be collected prospectively for 12 months and also a substantial amount of cycles will be analyzed retrospectively for the previous 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Péter Kovács, MD, Principal Investigator — Kaáli Institute, Budapest
Locations (1):
- Kaáli Institute, Budapest, Istenhegyi Út 54/A, Hungary